CLINICAL TRIAL: NCT07326917
Title: Effect of Learning Instruction Package on Patients' Knee Osteoarthritis Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Gamal Khairy Ali, Assistant lecturer of Medical - Surgical Nursing, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Instruction Package on Patient
Record Dates: First submitted 2025-12-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthristis

STUDY DESIGN:
Intervention Model Description: A quasi- experimental research design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- learning instruction package for improving Patients' Knee Osteoarthritis Outcomes (Experimental): participants in this group received learning instruction package
  Interventions: Behavioral: Learning Instruction Package

INTERVENTIONS:
Behavioral: Learning Instruction Package — participants received learning instruction package covered knowledge about knee osteoarthritis; definition, causes, risk factors, pathophysiology, signs, symptoms, and complications, and discussion how to improve knee osteoarthritis outcomes through weight management, diet management, regular exercise, application of compress, and how to apply it properly.

SUMMARY:
The aim of this study is to evaluate the effect of learning instruction package on patients' knee osteoarthritis outcomes.

DETAILED DESCRIPTION:
Musculoskeletal disorders are a group of diseases of the body's motor structures, particularly the bones, joints, muscles, fascia, and other supporting structures such as ligaments and cartilages. In fact, it is estimated that approximately 1.71 billion people are living with a musculoskeletal condition.

Osteoarthritis (OA) is the most common chronic joint disorder, characterized by local inflammation and joint structural change, it is associated with painful symptoms and loss of function leading to considerable impairment of quality of life. The rising rates of disability caused by osteoarthritis highlight the need for implementing preventative measures at early stages of the disease, which would especially benefit subjects at high risk for osteoarthritis development. Several joints are mainly affected by osteoarthritis, especially the knee, hip, hands, feet, shoulders, and spine.

Knee osteoarthritis (KOA) is a common chronic articular disease worldwide. It is also the most common form of osteoarthritis (OA) that affects the entire knee joint and is characterized by high morbidity and disability rates. It is ranked as the 10th largest contributor to global years lived with disabilities, and its prevalence has more than doubled in the last 10 years.

The main clinical symptoms of KOA are limb mobility difficulties, pain and swelling around the joint, which is more obvious after morning, and can lead to paralysis in the later stage. Pain is the key symptom of KOA and the main driver for functional disability and negative impact on different aspects of quality of life (QoL), including mobility, participation, mood and sleep. Patients may experience a serious impact on daily activities due to difficulty in walking, moving, climbing stairs, and while sitting on a chair with weakness of the thigh muscles.

Early diagnosis and treatment of knee osteoarthritis is more beneficial and easily managed compared to when it has worsened. The treatment includes nonpharmacological, pharmacological, and surgical modalities. Learning instruction has been recognized as one of the fundamental components for successful management of knee osteoarthritis, that involve teaching of patients regarding regular exercise, weight management, eating a balanced healthy diet, and applying of local cold or warm compress to improve patient knowledge, developing self-management and life skills.

Nurse plays a vital role in teaching and learning process, and providing valuable information for patients with knee osteoarthritis to improve health outcomes through modifying risk factors for disease progression, preventing further loss of function of the affected joints, relieving pain, improving joint function, optimizing daily living activities, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients.
* Age between 20 and 60 years.
* Clinically diagnosed with knee osteoarthritis.
* Able to communicate and follow instructions.

Exclusion Criteria:

* History of any orthopaedic surgical procedure on the affected knee.
* Presence of any physical disability that may interfere with participation.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Patients' Knee Osteoarthritis Outcomes | Basline, The first evaluation was conducted one month after completion of implementation of the learning instruction package, serving as a post-test, and the second evaluation was conducted one month after the first evaluation, as a follow-up.
  Assessment of patients' Knee Osteoarthritis Outcomes by using The Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire.
  The KOOS's five patient-relevant dimensions were scored separately: Pain (nine items), Symptoms (seven items), ADL Function (seventeen items), Sport and Recreation Function (five items), and Quality of Life (four items).

SECONDARY OUTCOMES:
Patients' knowledge regarding knee osteoarthritis questionnaire | Basline, The first evaluation was conducted one month after completion of implementation of the learning instruction package, serving as a post-test, and the second evaluation was conducted one month after the first evaluation, as a follow-up.
  Assessment of patients' knowledge about knee osteoarthritis pre & post learning instruction package.
  It included knowledge regarding disease and its management, that consisted of sixteen multiple-choice, closed-ended questions.
Body Mass Index (BMI) | Basline, The first evaluation was conducted one month after completion of implementation of the learning instruction package, serving as a post-test, and the second evaluation was conducted one month after the first evaluation, as a follow-up.
  BMI= Weight (kg) / Height (m2). It was categorized as follows: below 18.5 is underweight, 18.5- 24.9 is normal or healthy weight, 25- 29.9 is overweight, and 30 and above is obese.

CONTACTS AND LOCATIONS:
Overall Officials: Amany Mohammed Shebl, Professor, Study Director — Mansoura University; Wafaa Ismail Shereif, Professor, Study Director — Mansoura University
Locations (1):
- Faculty of Nursing. Mansoura University, Mansoura, Dakahlia 35516, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided